CLINICAL TRIAL: NCT05573672
Title: Dietary Counselling Plus Omega-3 Supplementation in the Treatment of Generalized Anxiety Disorder: A Randomized Wait-list Controlled Pilot Trial
Brief Title: Dietary Counselling Plus Omega-3 Supplementation in the Treatment of Generalized Anxiety Disorder
Acronym: EASe-GAD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: The Canadian College of Naturopathic Medicine (Other)
Collaborators: McGill University (Other); Netherlands Open University (Other); Massachusetts General Hospital (Other); Ekhagastiftelsen (Other); AquaOmega (Unknown); Lipid Analytical Laboratories Inc (Unknown); Mitacs (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CCNM_EASe-GADCT_2201v3
Record Dates: First submitted 2022-10-04; First posted 2022-10-10 (Actual); Results first posted 2025-04-04 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-03

CONDITIONS: Generalized Anxiety Disorder
Keywords: anxiety; generalized anxiety disorder; nutrition; diet; omega-3; lifestyle
MeSH Terms: conditions — Generalized Anxiety Disorder; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: This study will be wait-list controlled. Participants will be randomized to one of two groups. One group will begin the intervention immediately. The other will wait 12 weeks and then complete the intervention.
Who Masked: Outcomes Assessor
Masking Description: Collection of height and weight data will be completed by an individual blind to participant allocation. The statistician completing data analysis will be blind to allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Immediate Start (Experimental): Dietary Counselling (7 bi-weekly sessions) plus omega-3 supplementation
  Interventions: Combination Product: Dietary Counselling combined with Omega-3 Supplementation
- Waitlist Control (No Intervention): Participants will wait 12 weeks and then complete the same intervention as the Immediate Start arm.

INTERVENTIONS:
Combination Product: Dietary Counselling combined with Omega-3 Supplementation — Dietary Counselling: Seven, bi-weekly counselling sessions over 12-weeks conducted by a licensed Naturopathic Doctor. Each session will be 45-60 minutes in length. The recommendations will be based on the Mediterranean diet and the results of a recent scoping review which summarized the research related to diet and anxiety. The intervention will include motivational interviewing, mindful eating techniques, goal setting and action planning. A range of resources related to meal planning, recipes, cooking education, shopping lists and tracking sheets will be provided in an individualized manner.
  Dietary Supplement: AquaOmega High EPA Omega-3 capsules will be taken at a dose of four capsules, once daily (containing a total of 3456 mg of omega-3 fatty acids: 2659mg of Eicosapentaenoic acid (EPA), 532mg of docosahexaenoic acid (DHA), and 800IU of Vitamin D), with a meal.
  Arms: Immediate Start

SUMMARY:
This study will assess the feasibility and acceptability of a combination intervention including dietary counselling and omega-3 fatty acid supplementation among women with generalized anxiety disorder. It will be randomized and wait-list controlled with 25 participants completing the 12-week intervention immediately and the other 25 participants completing the intervention after a 12-week wait period.

DETAILED DESCRIPTION:
Generalized Anxiety Disorder (GAD) is a common mental health disorder involving high levels of worry or tension. The symptoms are persistent and distressing and interfere with an individual's functioning and quality of life. Clinical evidence suggests that nutritional interventions, based on the Mediterranean diet and omega-3 fatty acid supplementation improve the symptoms of depression. To date, the effect of diet change interventions on anxiety symptoms has not been studied in trials involving people with diagnosed anxiety disorders. The primary objective of this study is to test the feasibility and acceptability of a dietary counselling and omega-3 fatty acid supplementation intervention delivered to adult women with GAD. The secondary objectives include measuring changes in anxiety symptom severity, measuring changes in quality of life, measuring changes in biomarkers and evaluation of the components of the program.

This study is a randomized, wait-list controlled pilot trial delivering a 12-week, dietary counselling intervention and omega-3 supplementation to 50 adult women with GAD. Participant will complete seven individual counselling sessions which include nutrition education, personalized recommendations, mindful eating techniques, motivational interviewing, and goal setting. They will be provided with recipes, instructional videos, and food items. Questionnaires and blood work will be completed at baseline, after the wait period (for those in the wait-list group) and after the intervention. The questionnaires will measure changes in anxiety symptom severity, quality of life, diet quality, mindful eating behaviours, and self-efficacy and lab tests will measure changes in biomarkers of nutritional status. All participants will be asked to complete a brief satisfaction survey concerning the participant's level of satisfaction with the program, the aspects which were helpful or unhelpful, and opportunities for improvement. A sub-sample will be recruited to participate in a brief focus group in order to obtain more detailed qualitative responses about the participant experience and participant satisfaction. Additional information will be collected to characterize study participants including demographic information, body mass index, physical activity and food security.

Results from this study will lay the foundation for future large-scale studies in this area and may provide preliminary evidence of the role of diet counselling and omega-3 supplementation in the management of GAD.

ELIGIBILITY:
Inclusion Criteria:

* A person aged 18-65 years who currently identifies as a woman.
* Primary diagnosis of generalized anxiety disorder based on a clinical interview with a psychiatrist using the DSM-5 criteria.
* Moderate to severe anxiety as defined as a Beck Anxiety Inventory score of 22 or higher.
* Low quality diet as defined as a score of 8.5 or less on the MEDI-LITE tool.
* All psychiatric medication, psychotherapy and natural health products stable for the past four weeks.
* Established therapeutic relationship with a family doctor, psychiatrist, or clinical psychologist as their primary source of mental health care.
* Ability to swallow capsules.
* Ability to read in English and provide informed consent

Exclusion Criteria:

* Currently meets DSM-5 criteria for obsessive-compulsive disorder, bipolar disorder, a psychotic disorder, an eating disorder, or substance use disorder based on clinical interview with a psychiatrist.
* Current high level of suicidality assessed by trial psychiatrist using the Columbia Suicide Severity Scale.
* Starting or changing the dose of a psychiatric medication, psychotherapy, or natural health products in the past four weeks.
* Severe food allergies, intolerances or aversions that would prevent the individual from modifying their diet (includes aversion to bovine gelatin which is a component of the fish oil supplement).
* Current participation in a program, research study or treatment plan involving diet or lifestyle modification.
* Baseline Omega Score of >5% (suggesting adequacy of omega-3 fatty acids).
* Supplementation of greater than 4000IU of vitamin D daily for at least one month in the previous six months.
* Allergy to fish or any of the non-medicinal ingredients in the study product.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Participants who identify as women are eligible to participate
Enrollment: 50 (Actual)
Dates: Start 2022-08-12 (Actual); Primary Completion 2023-11-30 (Actual); Study Completion 2023-11-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Monique Aucoin, ND MSc, Principal Investigator — Canadian College of Naturopathic Medicine
Locations (1):
- Canadian College of Naturopathic Medicine, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Aucoin M, LaChance L, van der Wurff I, McLaren M, Monteiro S, Miller S, Jenkins A, Sabri E, Cooley K. Dietary counseling plus omega-3 supplementation in the treatment of generalized anxiety disorder: results of a randomized wait-list controlled pilot trial (the 'EASe-GAD Trial'). Nutr Neurosci. 2025 Jun;28(6):635-648. doi: 10.1080/1028415X.2024.2403901. Epub 2024 Sep 24. PMID 39316026
- [Derived] Aucoin M, LaChance L, van der Wurff I, Miller S, Naidoo U, Jenkins A, Cooley K. Dietary counselling plus omega-3 supplementation in the treatment of generalized anxiety disorder: protocol for a randomized wait-list controlled pilot trial (the "EASe-GAD Trial"). Pilot Feasibility Stud. 2023 Nov 10;9(1):186. doi: 10.1186/s40814-023-01414-y. PMID 37950301
- See also: Study Protocol — https://link.springer.com/article/10.1186/s40814-023-01414-y

RESULTS

PARTICIPANT FLOW:
Groups:
- Immediate Start: Dietary Counselling (7 bi-weekly sessions) plus omega-3 supplementation
  Dietary Counselling combined with Omega-3 Supplementation: Dietary Counselling: Seven, bi-weekly counselling sessions over 12-weeks conducted by a licensed Naturopathic Doctor. Each session will be 45-60 minutes in length. The recommendations will be based on the Mediterranean diet and the results of a recent scoping review which summarized the research related to diet and anxiety. The intervention will include motivational interviewing, mindful eating techniques, goal setting and action planning. A range of resources related to meal planning, recipes, cooking education, shopping lists and tracking sheets will be provided in an individualized manner.
  Dietary Supplement: AquaOmega High EPA Omega-3 capsules will be taken at a dose of four capsules, once daily (containing a total of 3456 mg of omega-3 fatty acids: 2659mg of Eicosapentaenoic acid (EPA), 532mg of docosahexaenoic acid (DHA), and 800IU of Vitamin D), with a meal.
Period: Overall Study
Arm/Group | Immediate Start | Waitlist Control
Started | 25 | 25
Completed | 23 | 23
Not Completed | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Immediate Start: began intervention immediately
- Waitlist: completed 12 week wait and then began intervention
- Total: Total of all reporting groups
Arm/Group | Immediate Start | Waitlist | Total
Number analyzed (Participants) | 24 | 25 | 49
Age, Continuous [Mean (Standard Deviation); unit: years] | 39 (14) | 35 (10) | 37 (12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 25 | 49
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black | 2 | 4 | 6
  East/Southeast Asian | 3 | 0 | 3
  First Nations/Indigenous/Metis | 1 | 0 | 1
  Latino | 2 | 1 | 3
  Middle Eastern | 1 | 0 | 1
  South Asian | 1 | 3 | 4
  White | 13 | 14 | 27
  Another race | 1 | 2 | 3
  Do not know | 0 | 1 | 1
Baseline Beck Anxiety Inventory Score [Mean (Standard Deviation); unit: units on a scale] | 26.2 (8.17) | 29.3 (11.71) | 27.8 (10.1)

OUTCOME MEASURES:

1. Primary Outcome: Feasibility of Participant Recruitment and Intervention Delivery
Description: Feasibility will be assessed by measuring the time to recruit and enrol 50 participants. Additionally, we will compare the intervention protocol with the intervention activities delivered.
Time Frame: 8 months
Population: 443 individuals contacted the study in 8 months. Of these, 50 met criteria for enrollment
Measure: Number; unit: months
Arm/Group | Immediate Start | Waitlist Control
Number analyzed (Participants) | 25 | 25
months | 8 | 8

2. Primary Outcome: Acceptability of the Intervention by Study Participants
Description: Acceptability will be assessed by measuring the number of diet counselling sessions completed. Additionally, participants will be asked to complete a brief satisfaction survey concerning the participant's level of satisfaction with the program, the aspects which were helpful or unhelpful, and opportunities for improvement. A sub-sample will be recruited to participate in a brief focus group in order to obtain more detailed qualitative responses about the participant experience and participant satisfaction.
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: number of sessions attended
Arm/Group | Immediate Start | Waitlist Control
Number analyzed (Participants) | 23 | 23
number of sessions attended | 6.4 (1.5) | 6.4 (1.9)

3. Secondary Outcome: Anxiety Symptom Severity: The Beck Anxiety Inventory
Description: The Beck Anxiety Inventory is a validated 21-item self-report inventory for measuring the severity of anxiety in participants with psychiatric illness. Answers to each item are given a score of 0 (not at all), 1 (mild), 2 (moderate) or 3 (severely), total scores range from 0 to 63 (minimal anxiety levels (0-7), mild anxiety (8-15), moderate anxiety (16-25), and severe anxiety (26-63)). The Beck Anxiety Inventory will be completed at baseline, after the wait period (for those in the waitlist group) and after the intervention.
Time Frame: 12 weeks
Population: Baseline questionnaires were completed by 24 participants in the immediate start group and 25 participants in the waitlist group. 23 participants in each group completed the 12 week questionnaires.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Immediate Start | Waitlist Control
Number analyzed (Participants) | 24 | 25
units on a scale
  Baseline | 26.2 [22.94 to 29.48] | 29.3 [24.73 to 33.91]
  12 weeks: number analyzed (Participants) | 23 | 23
  12 weeks | 11.0 [8.05 to 13.87] | 26.8 [22.09 to 31.56]

4. Secondary Outcome: Diet Quality: MEDI-LITE Questionnaire
Description: MEDI-LITE is a validated questionnaire that measures daily and weekly consumption of food typical and non-typical to the Mediterranean diet. Typical Mediterranean diet foods are scored 2 for high consumption, 1 more moderate and 0 for low. Non-typical Mediterranean diet foods are scored 2 for low consumption, 1 for moderate and 0 for high. Scores range from 0 (low consumption) to 18 (high consumption). The MEDI-LITE questionnaire will be completed to assess adherence to the Mediterranean diet at baseline, after the wait period (for those in the waitlist group) and after the intervention.
Time Frame: 12 weeks
Population: as for outcome 3
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Immediate Start | Waitlist Control
Number analyzed (Participants) | 24 | 25
score on a scale
  Baseline | 7.2 [6.32 to 8.10] | 7.1 [6.33 to 7.91]
  12 Weeks: number analyzed (Participants) | 23 | 23
  12 Weeks | 10.5 [9.55 to 11.49] | 6.9 [6.17 to 7.74]

5. Secondary Outcome: Quality of Life: PROMIS-29 v2.1
Description: The PROMIS-29 is a validated scale using 4 items scored on a 1-5 scale on intensity to assess 7 health domains (physical function, anxiety, depression, fatigue, sleep disturbance, ability to participate in social roles and activities and pain interference). Higher score equals more of the concept being measured (e.g., more Fatigue, more Physical Function). PROMIS-29 will be used to assess quality of life at baseline, after the wait period (for those in the waitlist group) and after the intervention.
Time Frame: 12 weeks
Population: as for outcome 3
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Immediate Start | Waitlist Control
Number analyzed (Participants) | 24 | 25
score on a scale
  physical, baseline | 4.54 [4.29 to 4.79] | 4.28 [3.93 to 4.63]
  physical, 12 weeks: number analyzed (Participants) | 23 | 23
  physical, 12 weeks | 4.79 [4.61 to 4.97] | 4.20 [3.82 to 4.56]
  anxiety, baseline | 3.42 [3.18 to 3.65] | 3.55 [3.29 to 3.81]
  anxiety, 12 weeks: number analyzed (Participants) | 23 | 23
  anxiety, 12 weeks | 2.16 [1.81 to 2.52] | 3.25 [2.92 to 3.58]
  depression, baseline | 2.59 [2.11 to 3.07] | 2.48 [2.03 to 2.95]
  depression, 12 weeks: number analyzed (Participants) | 23 | 23
  depression, 12 weeks | 1.72 [1.37 to 2.08] | 2.27 [1.83 to 2.72]
  fatigue, baseline | 3.78 [3.45 to 4.12] | 3.69 [3.35 to 4.03]
  fatigue, 12 weeks: number analyzed (Participants) | 23 | 23
  fatigue, 12 weeks | 2.75 [2.32 to 3.18] | 3.53 [3.09 to 9.97]
  social, baseline | 2.83 [2.38 to 3.28] | 2.81 [2.45 to 3.17]
  social, 12 weeks: number analyzed (Participants) | 23 | 23
  social, 12 weeks | 3.79 [3.31 to 4.28] | 3.14 [2.66 to 3.62]
  pain, baseline | 2.09 [1.59 to 2.59] | 2.24 [1.73 to 2.75]
  pain, 12 weeks: number analyzed (Participants) | 23 | 23
  pain, 12 weeks | 1.57 [1.19 to 1.96] | 2.14 [1.62 to 2.66]

6. Secondary Outcome: Mindful Eating Behaviour: Mindful Eating Questionnaire
Description: The MEQ is a 28-item scale that measures five factors associated with mindful eating (emotional responses, distraction, external cues, awareness and disinhibition). The questionnaire will be used to measure behaviour change and qualitatively assess the acceptability of the intervention. Each item is scored on a 1-4 scale, higher scores signify more mindful eating. The scores are added together and divided by the number of items answered to get a total summary score. The minimum score is 1 and the maximum score is 4. The MEQ will be completed at baseline, after the wait period (for those in the waitlist group) and after the intervention.
Time Frame: 12 weeks
Population: as for outcome 3
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Immediate Start | Waitlist Control
Number analyzed (Participants) | 24 | 25
units on a scale
  MEQ, baseline | 2.5 [2.38 to 2.73] | 2.6 [2.46 to 2.77]
  MEQ, 12 weeks: number analyzed (Participants) | 23 | 23
  MEQ, 12 weeks | 2.88 [2.73 to 3.03] | 2.5 [2.37 to 2.69]

7. Secondary Outcome: Self Efficacy: General Self-Efficacy Scale
Description: The GSE is a 10-item validated questionnaire that measures an individual's belief in their ability to overcome and respond to difficult scenarios. Answers to each item are given a score of 0 (not at all true), 1 (barely true), 3 (moderately true) or 4 (exactly true), higher scores correlate to greater self-efficacy. The minimum score is 10 and the maximum score is 40. The GSE will be completed at baseline, after the wait period (for those in the waitlist group) and after the intervention.
Time Frame: 12 weeks
Population: as for outcome 3
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Immediate Start | Waitlist Control
Number analyzed (Participants) | 24 | 25
units on a scale
  GSE, baseline | 28.9 [27.24 to 30.59] | 28.2 [26.20 to 30.20]
  GSE, 12 weeks: number analyzed (Participants) | 23 | 23
  GSE, 12 weeks | 32.3 [30.70 to 33.91] | 28.2 [26.49 to 29.95]

8. Secondary Outcome: OmegaScore
Description: Summed EPA, DHA and DPA as a percentage of total fatty acids in whole blood as a measure of omega-3 status. This blood test will be completed at baseline, after the wait period (for those in the waitlist group) and after the intervention.
Time Frame: 12 weeks
Population: all 50 participants assessed at baseline. 21 and 23 assessed at 12 weeks
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | Immediate Start | Waitlist Control
Number analyzed (Participants) | 25 | 25
percentage
  baseline | 3.58 (0.74) | 3.43 (0.50)
  week 12: number analyzed (Participants) | 21 | 23
  week 12 | 7.18 (2.12) | 3.47 (0.92)

9. Secondary Outcome: Fasting Cholesterol Panel
Description: Measures of serum cholesterol including LDL, HDL, triglycerides and total cholesterol. This blood test will be completed at baseline, after the wait period (for those in the waitlist group) and after the intervention.
Time Frame: 12 weeks
Population: at 12 weeks, data were collected for 21 in the immediate start group and 22 in the waitlist group
Measure: Mean (95% Confidence Interval); unit: mmol/L
Arm/Group | Immediate Start | Waitlist Control
Number analyzed (Participants) | 24 | 23
mmol/L
  triglycerides, baseline | 1.13 [0.93 to 1.32] | 1.02 [0.89 to 1.15]
  triglycerides, week 12: number analyzed (Participants) | 21 | 22
  triglycerides, week 12 | 0.88 [0.69 to 1.06] | 0.88 [0.74 to 1.03]
  Total cholesterol, baseline | 4.72 [4.24 to 5.19] | 4.80 [4.30 to 5.30]
  Total cholesterol, week 12: number analyzed (Participants) | 21 | 22
  Total cholesterol, week 12 | 4.62 [4.11 to 5.13] | 4.75 [4.32 to 5.18]
  LDL, baseline | 2.63 [2.20 to 3.05] | 2.84 [2.42 to 3.74]
  LDL, week 12: number analyzed (Participants) | 21 | 22
  LDL, week 12 | 2.67 [2.21 to 3.57] | 2.86 [2.50 to 3.21]
  HDL, baseline | 1.58 [1.40 to 1.75] | 1.50 [1.34 to 1.66]
  HDL, week 12: number analyzed (Participants) | 21 | 22
  HDL, week 12 | 1.55 [1.37 to 1.73] | 1.49 [1.32 to 1.67]

10. Secondary Outcome: Hemoglobin A1c
Description: Measure of the average blood sugar in the past 3 months. This blood test will be completed at baseline, after the wait period (for those in the waitlist group) and after the intervention.
Time Frame: 12 weeks
Population: at 12 weeks, data were collected for 21 in the immediate start group and 22 in the waitlist group
Measure: Mean (95% Confidence Interval); unit: percentage
Arm/Group | Immediate Start | Waitlist Control
Number analyzed (Participants) | 24 | 23
percentage
  baseline | 5.35 [5.23 to 5.46] | 5.52 [5.15 to 5.88]
  12 weeks: number analyzed (Participants) | 21 | 22
  12 weeks | 5.36 [5.24 to 5.48] | 5.57 [5.16 to 5.97]

11. Secondary Outcome: Serum Vitamin C
Description: Measure of serum levels of vitamin C as an objective marker for fruit and vegetable intake. This blood test will be completed at baseline, after the wait period (for those in the waitlist group) and after the intervention.
Time Frame: 12 weeks
Population: at 12 weeks, data were collected for 21 in the immediate start group and 22 in the waitlist group
Measure: Mean (95% Confidence Interval); unit: umol/L
Arm/Group | Immediate Start | Waitlist Control
Number analyzed (Participants) | 24 | 23
umol/L
  baseline | 49.00 [41.55 to 56.45] | 41.36 [33.99 to 48.74]
  week 12: number analyzed (Participants) | 21 | 22
  week 12 | 50.90 [43.17 to 58.64] | 42.25 [35.24 to 49.26]

12. Secondary Outcome: Serum Beta-carotene
Description: Measure of serum levels of beta-carotene as an objective marker for fruit and vegetable. This blood test will be completed at baseline, after the wait period (for those in the waitlist group) and after the intervention.
Time Frame: 12 weeks
Population: at 12 weeks, data were collected for 21 in the immediate start group and 22 in the waitlist group
Measure: Mean (95% Confidence Interval); unit: umol/L
Arm/Group | Immediate Start | Waitlist Control
Number analyzed (Participants) | 24 | 23
umol/L
  baseline | 0.53 [0.38 to 0.67] | 0.40 [0.29 to 0.52]
  week 12: number analyzed (Participants) | 21 | 22
  week 12 | 0.66 [0.49 to 0.83] | 0.44 [0.32 to 0.57]

13. Secondary Outcome: C-reactive Protein
Description: CRP will be used to measure inflammation levels. This blood test will be completed at baseline, after the wait period (for those in the waitlist group) and after the intervention.
Time Frame: 12 weeks
Population: at 12 weeks, data were collected for 21 in the immediate start group and 22 in the waitlist group
Measure: Mean (95% Confidence Interval); unit: mg/L
Arm/Group | Immediate Start | Waitlist Control
Number analyzed (Participants) | 24 | 23
mg/L
  baseline | 3.11 [1.97 to 4.26] | 6.60 [2.77 to 10.43]
  week 12: number analyzed (Participants) | 21 | 22
  week 12 | 4.06 [2.27 to 5.85] | 7.49 [2.78 to 12.19]

14. Secondary Outcome: HOMA-IR
Description: Homeostatic Model Assessment of Insulin Resistance, calculated using fasting insulin and fasting glucose. Formula: fasting glucose (mg/dL) X fasting insulin (mU/L) / 405. A higher value suggests more insulin resistance. These blood tests and calculation will be completed at baseline, after the wait period (for those in the waitlist group) and after the intervention.
Time Frame: 12 weeks
Population: at 12 weeks, data were collected for 21 in the immediate start group and 22 in the waitlist group
Measure: Mean (95% Confidence Interval); unit: HOMA-IR index
Arm/Group | Immediate Start | Waitlist Control
Number analyzed (Participants) | 24 | 23
HOMA-IR index
  baseline | 2.94 [2.01 to 3.87] | 4.05 [1.86 to 6.25]
  12 weeks: number analyzed (Participants) | 21 | 22
  12 weeks | 2.92 [1.89 to 3.95] | 4.81 [0.93 to 8.69]

ADVERSE EVENTS:
Time Frame: 12 weeks
Arm/Group | Immediate Start | Waitlist Control
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/25
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/25
Other Adverse Events (participants affected / at risk) | 21/25 | 0/25
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Immediate Start (N=25) | Waitlist Control (N=25)
GI symptoms (Gastrointestinal disorders) | 19 (19) | 0 — belching (n=5), diarrhea (n=5), gastroesophageal reflux (n=3), bloating (n=3), nausea (n=2) and constipation (n=1)
heart palpitations (Cardiac disorders) | 2 (2) | 0 (0)
pruritis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-11-10): https://cdn.clinicaltrials.gov/large-docs/72/NCT05573672/Prot_SAP_001.pdf
  • Informed Consent Form (2023-01-05): https://cdn.clinicaltrials.gov/large-docs/72/NCT05573672/ICF_002.pdf